CLINICAL TRIAL: NCT06718023
Title: Effect of Diverse Training Programs on Prevention of Sarcopenia in Postmenopausal Women
Brief Title: Diverse Training Programs and Sarcopenia in Postmenopausal Women
Acronym: PA&SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AWFiS/2023_7_ZO; without grant number (Other Grant/Funding Number: Gdansk University of Physical Education and Sport)
Record Dates: First submitted 2024-10-29; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Sarcopenia
Keywords: sarcopenia; postmenopausal women; Nordic walking; Strength training; Bungy Pump Exercises
MeSH Terms: conditions — Sarcopenia | interventions — Nordic Walking; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nordic walking (Experimental): Training is about 60 minutes each time, 3 times a week, each interval of 1 or 2 days, a total of 12 weeks. The primary focus is on utilizing a specialized pole for engaging in cross-country walking. This regimen entails approximately 10 minutes of warm-up exercises, followed by around 40 minutes of brisk walking, and concluding with a period of relaxation stretching lasting between 5 to 8 minutes.
  Interventions: Behavioral: Nordic walking
- Daily life (No Intervention): The individuals engaged in routine daily tasks, while being advised against incorporating any supplementary physical exertion.
- Strength training (Experimental): Strength training was conducted in the gym with progressively increasing resistance from 65% to 75% of the maximum weight (one-repetition maximum (1-RM)). Participants performed 10-13 repetitions of the exercise in one serie. The training was carried out in station form and consisted of 10-13 exercises. There were rest intervals of 60-90 seconds between exercises. As intended, the training was comprehensive, i.e. it affected the muscles of the arms, legs, torso, abdomen and chest.
  Interventions: Behavioral: Strength training
- Bungy Pump Exercises (Experimental): The training lasts approximately 60 minutes each time, 3 times a week, for a period of 12 weeks. The main emphasis is placed on the use of a specialist Bungy Pump pole. Bungy Pump training allows participants to combine aerobic and strength training. Bungy Pump poles contain a built-in shock absorber (RSA) in the form of an elastic band. The additional resistance generated by the stretched band increases the overall intensity of the exercise and increases calorie consumption. The program classes will include approximately 10 minutes of warm-up exercises, followed by approximately 40 minutes of brisk walking, and at the end a period of relaxation stretching lasting from 5 to 8 minutes.
  Interventions: Behavioral: Bungy Pump Exercises

INTERVENTIONS:
Behavioral: Nordic walking — NW training sessions are conducted by a certified NW instructor leading participants in the outdoor forest of Gdansk. Training is about 60 minutes each time, 3 times a week, each interval of 1 or 2 days, a total of 12 weeks. Participants used professional Nordic Pole.
  Arms: Nordic walking
Behavioral: Strength training — Strength training was conducted in the gym with progressively increasing resistance from 65% to 75% of the maximum weight (one-repetition maximum (1-RM)). Participants performed 10-13 repetitions of the exercise in one serie. The training was carried out in station form and consisted of 10-13 exercises. There were rest intervals of 60-90 seconds between exercises. As intended, the training was comprehensive, i.e. it affected the muscles of the arms, legs, torso, abdomen and chest.
  Arms: Strength training
Behavioral: Bungy Pump Exercises — Buny Pump training sessions are conducted by a certified BP instructor leading participants in the outdoor forest of Gdansk. Training is about 60 minutes each time, 3 times a week, , a total of 12 weeks. Participants used professional Bungy Pump Pole.
  Arms: Bungy Pump Exercises

SUMMARY:
This study explored preventive measures for sarcopenia in apparently healthy postmenopausal women. The investigators implemented a short Nordic walking intervention, Bungy Pumo exercises and strength training, and conducted a 3-month training program as an intervention method. The subjects divided into the NW (Nordic walking) test group, the ST (Strength Training) test group, BP (Bungy Pump exercises) test group and the control group, which engaged in regular daily activities without any additional physical exercise. The collected experimental data then processed and analyzed to objectively assess the benefits and limitations of different interventions.

DETAILED DESCRIPTION:
The tests were conducted twice (before and after the training period). Each test lasted two days and will be preceded by a 7-day measurement of physical activity using sport testers. On the first day, blood tests, microbiota, body composition and a preliminary analysis of diet diaries were performed. On the second day, physical fitness tests were carried out in the Physical Exercise Laboratory of the AWFiS in Gdańsk. Biological material (blood serum and feces) was frozen for testing by the project contractors in the Laboratory of Genetics in Sports of the AWFiS. The subjects were required to keep a diet diary in which they recorded meals during the 3 days preceding the blood and intestinal microbiota test.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women over 60 years old (i.e. more than 12 months since their last menstrual cycle).

There were no contraindications to exercise after case reports and initial diagnosis.

Informed consent must be signed, agreeing to participate in research and physical exercise programs.

Exclusion Criteria:

Uncontrolled high blood pressure. Coronary artery disease. Rheumatoid arthritis. Type 2 diabetes. Respiratory diseases and lung diseases. Are taking or have used antibiotics and/or antifungal therapy in the past 4 weeks.

Unwillingness to stick to a prescribed schedule.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle index | From enrollment to the end of treatment at 2 weeks
  SMI in InBody is calculated as follows: SMI= sum of segmental muscle mass (two arms and two legs) ÷ height 2
Gait Speed | From enrollment to the end of treatment at 2 weeks
  In order to harmonize the pace measurement method, the 2019 Asian Sarcopenia Working Group recommends the time it takes to walk 6 meters at a normal pace from moving as a measure of average pace. The test is carried out in an inspection room that is more than 8 meters long. Crutches that participants normally use can also be used. The start and end of the 6-meter distance are clearly marked. Subjects stand with their toes touching the starting line, and after being instructed to move forward at their usual speed, subjects start walking, inspectors start timing, and when subjects fully cross the 6-meter mark with one foot, inspectors stop timing. The test is performed twice, recording the shortest time (in seconds) required to complete each distance. The smaller the value, the faster the walking speed, the better the physical ability.
Hand Strength | From enrollment to the end of treatment at 2 weeks
  HS was measured to estimate muscle strength and was performed with a hand dynamometer (SAEHAN Digital Hand Dynamometer, SAEHAN, Changwon, Korea). During the HS test, participants had to hold the dynamometer in their hand with the arm stretched parallel to the body while being instructed to stand upright. This measure was performed three times on the dominant hand with a rest interval of 1 min between measurements; finally, the best performance was used as the maximum peak (PK) of HS (in kg). The statistical analysis also included mean peak (mean PK).The higher the grip strength value, the greater the muscle strength, the better the physical ability.
Skeletal Muscle Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes.The higher the number, the more muscle the human body has.The ideal skeletal muscle content for men is 47% of standard body weight and 42% of standard body weight for women. A 10% move up or down is considered normal.

SECONDARY OUTCOMES:
Right Arm Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher number indicates more muscle in the right arm.
Left Arm Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher number indicates more muscle in the left arm.
Trunk Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher number indicates more muscle in the trunk.
Right Leg Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher number indicates more muscle in the right leg.
Left Leg Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher number indicates more muscle in the left leg.
Skeletal Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The calculation method of SLM is different from that of SMM. The SLM in InBody report paper is the sum of protein, body water, and extracosseous inorganic salts. The ideal SLM for men is 80% of standard body weight and 72% of standard body weight for women. A 10% move up or down is considered normal.
PEAK AWY | From enrollment to the end of treatment at 2 weeks
  Peak knee extension muscle strength.Using Biodex System 4 Pro™ dynamometers (Biodex Medical Systems, Inc.) Data collection using Compaq Desk Pro personal computers and Biodex software, using the Biodex standard protocol. After a standardized warm-up, the subject is positioned in the equipment as required by the manufacturer's manual (sitting position, arms hanging down along the body, hands holding the outside handle, torso, buttocks and subject thighs secured by straps, knee flexion to 90°). The test uses the scheme reported by Symons et al., with some modifications. The isometric muscle strength test was performed using three maximum contractions, each lasting 5 seconds with an interval of 30 seconds. Adjust the seat position according to the length of each subject's legs. Data were analyzed using the results of the dominant lower limbs.
  The greater the value of this index, the stronger the isometric contraction force of the knee extensor muscle.
PEAK TWD | From enrollment to the end of treatment at 2 weeks
  Peak knee flexor strength. Using Biodex System 4 Pro™ dynamometers (Biodex Medical Systems, Inc.) Data collection using Compaq Desk Pro personal computers and Biodex software, using the Biodex standard protocol. After a standardized warm-up, the subject is positioned in the equipment as required by the manufacturer's manual (sitting position, arms hanging down along the body, hands holding the outside handle, torso, buttocks and subject thighs secured by straps, knee flexion to 90°). The test uses the scheme reported by Symons et al., with some modifications. The isometric muscle strength test was performed using three maximum contractions, each lasting 5 seconds with an interval of 30 seconds. Adjust the seat position according to the length of each subject's legs. Data were analyzed using the results of the dominant lower limbs.
  The higher the value of this index, the stronger the isometric contraction force of knee flexor muscle.
Arm Circumference | From enrollment to the end of treatment at 2 weeks
  A tape measure was used to directly measure the circumference of the left and right upper arms of the participants. The larger the value of the index, the larger the arm circumference, but it can only be used as a reference indicator and cannot specifically evaluate the physical function
ChairStand | From enrollment to the end of treatment at 2 weeks
  The participants stood up as fast as they could on a chair of suitable height for 30 seconds. The greater the value of this test, the more times it is proved to be completed, and the lower limb muscle strength can be indirectly evaluated.
ArmCurl | From enrollment to the end of treatment at 2 weeks
  Participants were asked to sit in a chair holding a 2KG weight with one arm and complete the maximum number of arm curls within 30 seconds. The greater the number of bends, the better the upper body strength may prove.
TUG | From enrollment to the end of treatment at 2 weeks
  Time up and go.The TUG test measures the time(s) required for a subject to rise from a chair, walk 3 m, turn around, walk back to the chair, and sit down. It has been shown to be a predictor of sarcopenia in hospitalized patients with a mean age of 70.4±7.7 years.The smaller the value, the shorter the completion time, and the better the physical function.
TandemBalance | From enrollment to the end of treatment at 2 weeks
  Participants used the "toe" stick to the "heel" in a straight line walking way, with the fastest speed to complete 2 meters. The smaller the value, the faster the walking speed, which may represent better balance ability.
Muscle Strength Indices | From enrollment to the end of treatment at 2 weeks
  The index includes 2 upper limb muscle strength indexes and 2 lower limb muscle strength indexes, and the formula is as follows:
  1. HS/BM
  2. HS/BMI
  3. Knee extensor strength /BM
  4. Knee flexor strength /BM A higher value for this indicator may mean greater muscle strength.
Myostatin | From enrollment to the end of treatment at 3 months
  Myostatin is a protein whose units are the same as those of other proteins, usually expressed in moles (mol/L).
  The MAGPIX platform enables multiplex tests, which allow for multi-parameter detection of several to several dozen analytes in a single sample of small volume (~40ul). The MAGPIX (xMAP®) system is based on the principles of the ELISA test and uses the technology of paramagnetic microspheres coated with antibodies. One panel allows for simultaneous determination of several to several dozen markers in each sample. ELISA (enzyme-linked immunosorbent assay) is an immunoenzymatic test used to detect and quantify proteins contained in the tested sample, such as antibodies or protein antigens. The ELISA technique is widely used in biomedical research, both scientific and diagnostic. It is a fast, accurate and easy to perform method. Consumables: nitrile gloves, pipette tips 10-200ul, pipette tips 100-1000ul, eppendorff tubes, other (falcon tubes, lignin, etc.).
Irisin | From enrollment to the end of treatment at 3 months.
  The unit of irisin is molecular weight and its value is 298.25.
  The MAGPIX platform enables multiplex tests, which allow for multi-parameter detection of several to several dozen analytes in a single sample of small volume (~40ul). The MAGPIX (xMAP®) system is based on the principles of the ELISA test and uses the technology of paramagnetic microspheres coated with antibodies. One panel allows for simultaneous determination of several to several dozen markers in each sample. ELISA (enzyme-linked immunosorbent assay) is an immunoenzymatic test used to detect and quantify proteins contained in the tested sample, such as antibodies or protein antigens. The ELISA technique is widely used in biomedical research, both scientific and diagnostic. It is a fast, accurate and easy to perform method. Consumables: nitrile gloves, pipette tips 10-200ul, pipette tips 100-1000ul, eppendorff tubes, other (falcon tubes, lignin, etc.).
BDNF | From enrollment to the end of treatment at 3 months.
  BDNF (brain-derived neurotrophic factor) assay unit is mainly pg/mL.
  The MAGPIX platform enables multiplex tests, which allow for multi-parameter detection of several to several dozen analytes in a single sample of small volume (~40ul). The MAGPIX (xMAP®) system is based on the principles of the ELISA test and uses the technology of paramagnetic microspheres coated with antibodies. One panel allows for simultaneous determination of several to several dozen markers in each sample. ELISA (enzyme-linked immunosorbent assay) is an immunoenzymatic test used to detect and quantify proteins contained in the tested sample, such as antibodies or protein antigens. The ELISA technique is widely used in biomedical research, both scientific and diagnostic. It is a fast, accurate and easy to perform method. Consumables: nitrile gloves, pipette tips 10-200ul, pipette tips 100-1000ul, eppendorff tubes, other (falcon tubes, lignin, etc.).

OTHER OUTCOMES:
Creatinine | From enrollment to the end of treatment at 2 weeks
  creatinine [mg/dl]. In all measurements, the mean value of the measurement in the tested group and the standard deviation of the results will be reported.
  After obtaining blood samples from participants in the blood laboratory, investigators performed blood biomarker analysis using the Luminex method. Studies have shown that creatinine and creatine kinase are significantly reduced in patients with sarcopenia. Therefore, they were used as part of the results measurement in this study.
Creatine kinase | From enrollment to the end of treatment at 2 weeks
  creatine kinase [U/l]. In all measurements, the mean value of the measurement in the tested group and the standard deviation of the results will be reported.
  After obtaining blood samples from participants in the blood laboratory, investigators performed blood biomarker analysis using the Luminex method. Studies have shown that creatinine and creatine kinase are significantly reduced in patients with sarcopenia. Therefore, they were used as part of the results measurement in this study.
Body Fat Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes.The higher the value of this index, the higher the body fat content.
Fat-Free Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The higher the value of this index, the heavier the body weight without fat.
BMI | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 720 analyzer (Biospace, Seoul, Korea), participants wore light clothing and no shoes. The average person's BMI is usually between 18 and 23.
Microbiome analysis | From enrollment to the end of treatment at 3 months
  The microbiome test will be performed at the AWFiS Sports Genetics Laboratory. DNA will be isolated using a Bead Ruptor 24 Elite homogenizer and QIAamp PowerFecal Pro DNA Kits (Qiagen) according to the manufacturer's procedure. The quality and quantity of the isolated material will be checked on a NanoDrop 1000 spectrophotometer (Thermo Scientific), Qubit 4.0 fluorometer (ThermoFisher). Sequencing in PE mode (2x150 bp) will be performed on the NovaSeq platform (Illumina). Data analysis will be performed using a specially created pipeline based on several programs such as: MG-RAST, Mothur or CLUSTOM, R program, etc.
CRP | From enrollment to the end of treatment at 3 months
  CRP is an acute phase reaction protein, the unit of CRP is: mg/L. Blood collection and C-reactive protein assay will be performed by an external company.
IL-6 | From enrollment to the end of treatment at 3 months.
  The unit of IL-6 (interleukin-6) is (pg/mL).
  Fasting venous blood samples will be collected after a minimum of 12 hours overnight. Blood will be collected in Sarstedt S-Monovette tubes without anticoagulants but with the addition of coagulation factors to obtain serum. Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Levels of inflammatory markers CRP, IL-6 and TNF-alpha will be determined using the MAGPIX fluorescence detection system (Luminex Corp., Austin, TX, USA) and the Luminex Human Magnetic Assay 6-Plex according to the manufacturer's protocols. Data acquisition and analysis will be performed using xPONENT software and Quantist Luminex by Bio-Techne (Luminex Corp., Austin, TX, USA).
TNF-α | From enrollment to the end of treatment at 3 months.
  TNF-α (tumor necrosis factor-α) has two molecular weights: 17kD monomer form and 51kD trimer form . According to the molecular weight, the concentration unit of TNF-α can be converted. For example, in the monomer form of TNF-α, 1ug is approximately equal to 0.06nmol; In trimer form TNF-α, 1ug is equal to approximately 0.02nmol .
  Serum samples will be processed according to standard laboratory procedures, aliquoted and stored at -80°C until analysis. Levels of inflammatory markers CRP, IL-6 and TNF-alpha will be determined using the MAGPIX fluorescence detection system (Luminex Corp., Austin, TX, USA) and the Luminex Human Magnetic Assay 6-Plex according to the manufacturer's protocols. Data acquisition and analysis will be performed using xPONENT software and Quantist Luminex by Bio-Techne (Luminex Corp., Austin, TX, USA).
Nutrition assessment | From enrollment to the end of treatment at 3 months
  Nutrition analysis (nutrient and caloric content) based on diet diaries kept by the study participants using diet analysis software.
  Nutritional analysis in the Nuvero program is based on entering data from diet diaries and assessing the consumption of basic nutrients and caloric content in the context of the nutritional needs of the person being examined. The process begins with collecting detailed information about the products and dishes consumed, which are recorded in the diet diaries kept by the person being examined. This information should include: the type of products consumed, the size of portions and the method of their preparation.
  The collected data is entered into the Nuvero program, selecting from the available database the products and dishes that most closely correspond to the entries in the diary. If necessary, modifications to the ingredients or methods of preparing dishes should be taken into account to ensure the accuracy of the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Ossowski Professor, PHD, Principal Investigator — AKADEMIA WYCHOWANIA FIZYCZNEGO I SPORTU
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided
There are some privacy concerns

REFERENCES:
- [Background] Ossowski ZM, Skrobot W, Aschenbrenner P, Cesnaitiene VJ, Smaruj M. Effects of short-term Nordic walking training on sarcopenia-related parameters in women with low bone mass: a preliminary study. Clin Interv Aging. 2016 Nov 30;11:1763-1771. doi: 10.2147/CIA.S118995. eCollection 2016. PMID 27942207
- [Background] Li T, Yin D, Shi R. Gut-muscle axis mechanism of exercise prevention of sarcopenia. Front Nutr. 2024 Aug 16;11:1418778. doi: 10.3389/fnut.2024.1418778. eCollection 2024. PMID 39221163
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Gorbatov SY, Aksenova EI, Burkovskaya YV, Ivanov AV, Gazheva AV. [Global demographic problem and active aging (literature review)]. Probl Sotsialnoi Gig Zdravookhranenniiai Istor Med. 2023 Oct;31(Special Issue 2):1109-1114. doi: 10.32687/0869-866X-2023-31-s2-1109-1114. Russian. PMID 38069871
- [Background] Christensen K, Doblhammer G, Rau R, Vaupel JW. Ageing populations: the challenges ahead. Lancet. 2009 Oct 3;374(9696):1196-208. doi: 10.1016/S0140-6736(09)61460-4. PMID 19801098
- [Background] Partridge L, Deelen J, Slagboom PE. Facing up to the global challenges of ageing. Nature. 2018 Sep;561(7721):45-56. doi: 10.1038/s41586-018-0457-8. Epub 2018 Sep 5. PMID 30185958